CLINICAL TRIAL: NCT07225517
Title: A Phase 1, Randomized, Blinded, Placebo-Controlled, Single- and Multiple-Ascending-Dose Study to Investigate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of BIIB145 in Healthy Adult Participants
Brief Title: A Study to Learn More About the Safety of BIIB145 and How it is Processed in the Body of Healthy Adult Participants
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Biogen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 302HV101
Record Dates: First submitted 2025-11-04; First posted 2025-11-06 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Healthy Volunteer

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (12):
- Part A [Single Ascending Dose (SAD)]: BIIB145 Cohort 1A (Experimental): Participants will receive Dose A of BIIB145 or a matching placebo on Day 1 in a fasted state.
  Interventions: Drug: BIIB145; Drug: Placebo
- Part A (SAD): BIIB145 Cohort 2A (Experimental): Participants will receive Dose B of BIIB145 or a matching placebo on Day 1 in a fasted state.
  Interventions: Drug: BIIB145; Drug: Placebo
- Part A (SAD): BIIB145 Cohort 3A (Experimental): Participants will receive Dose C of BIIB145 or a matching placebo on Day 1 in a fasted state.
  Interventions: Drug: BIIB145; Drug: Placebo
- Part A (SAD): BIIB145 Cohort 4A (Experimental): Participants will receive Dose D of BIIB145 or a matching placebo on Day 1 in a fasted state.
  Interventions: Drug: BIIB145; Drug: Placebo
- Part A (SAD): BIIB145 Cohort 5A (Experimental): Participants will receive Dose E of BIIB145 or a matching placebo on Day 1 in a fasted state.
  Interventions: Drug: BIIB145; Drug: Placebo
- Part A (SAD): BIIB145 Cohort 6A (Experimental): Participants will receive Dose F of BIIB145 or a matching placebo on Day 1 in a fasted state.
  Interventions: Drug: BIIB145; Drug: Placebo
- Part A (SAD): BIIB145 Cohort 7A (Experimental): Participants will receive Dose G of BIIB145 or a matching placebo on Day 1 in a fasted state.
  Interventions: Drug: BIIB145; Drug: Placebo
- Part B [Food Effect]: BIIB145 Cohort 1B (Experimental): Participants will receive BIIB145 on Day 1 in the fasted state, followed by the fed state in the first sequence, and vice versa in the second sequence. A washout period of 7 days will be maintained between the two sequences. Dose will be determined based on safety and PK data of SAD Cohort 6A as well as safety, PK and pharmacodynamics (PD) data from previous cohorts.
  Interventions: Drug: BIIB145
- Part C [Multiple Ascending Dose (MAD)]: BIIB145 Cohort 1C (Experimental): Participants will receive Dose B of BIIB145 or a matching placebo administered orally once daily for 14 days in a fasted state.
  Interventions: Drug: BIIB145; Drug: Placebo
- Part C [Multiple Ascending Dose (MAD)]: BIIB145 Cohort 2C (Experimental): Participants will receive Dose C of BIIB145 or a matching placebo administered orally once daily for 14 days in a fasted state.
  Interventions: Drug: BIIB145; Drug: Placebo
- Part C [Multiple Ascending Dose (MAD)]: BIIB145 Cohort 3C (Experimental): Participants will receive Dose H of BIIB145 or a matching placebo administered orally once daily for 14 days in a fasted state.
  Interventions: Drug: BIIB145; Drug: Placebo
- Part C [Multiple Ascending Dose (MAD)]: BIIB145 Cohort 4C (Experimental): Participants will receive Dose F of BIIB145 or a matching placebo administered orally once daily for 14 days in a fasted state.
  Interventions: Drug: BIIB145; Drug: Placebo

INTERVENTIONS:
Drug: BIIB145 — Administered orally
Drug: Placebo — Administered orally
  Arms: Part A (SAD): BIIB145 Cohort 2A; Part A (SAD): BIIB145 Cohort 3A; Part A (SAD): BIIB145 Cohort 4A; Part A (SAD): BIIB145 Cohort 5A; Part A (SAD): BIIB145 Cohort 6A; Part A (SAD): BIIB145 Cohort 7A; Part A [Single Ascending Dose (SAD)]: BIIB145 Cohort 1A; Part C [Multiple Ascending Dose (MAD)]: BIIB145 Cohort 1C; Part C [Multiple Ascending Dose (MAD)]: BIIB145 Cohort 2C; Part C [Multiple Ascending Dose (MAD)]: BIIB145 Cohort 3C; Part C [Multiple Ascending Dose (MAD)]: BIIB145 Cohort 4C

SUMMARY:
In this study, researchers will learn for the first time about the safety of a study drug called BIIB145 and how the body responds to it. This is a "Phase 1" study. This kind of study is an early step in clinical research where the goal is to focus on the safety of the study drug. Another goal may be to learn how the study drug is processed by the body. BIIB145 was designed to help people with multiple sclerosis (MS). But, before it can be tested in people with MS, it must first be tested in healthy volunteers to learn about its safety and other effects.

The main goal of this study is to learn about the safety of BIIB145 and how it is processed by the body, with or without food.

The main questions researchers want to answer are:

* How many participants have adverse events and serious adverse events during the study? An adverse event is a health problem that may or may not be caused by the study drug.
* How does BIIB145 affect the participants' overall health?

Researchers will also learn more about:

* How BIIB145 is processed by the body, with or without food.

This study will be done as follows:

* Participants will be screened to check if they can join the study. The screening period will be up to 28 days, after which participants will check into the study research center.
* There will be 3 parts to this study.
* Part 1: Participants will take a single dose of BIIB145 or a placebo after not eating overnight. A placebo is something that looks like the study drug but does not contain any medicine. A placebo is also given in the same way as the study drug. Participants in Part 1 will be in the study for up to 42 days.
* Part 2: This part of the study will have a "crossover" design. This means that all participants in Part 2 will all take BIIB145 twice, once with food and once without food. When taken with food, they will finish a meal about 30 minutes before their dose. Without food, they will not eat overnight before taking their dose. But, the order in which they take BIIB145 with or without food depends on the group to which they are randomly assigned. Participants in Part 2 will be in the study for up to 56 days.
* Part 3: Participants will take a dose of BIIB145 or the placebo once a day for 14 days. For each dose, participants will not eat overnight before taking it. Participants in Part 3 will be in the study for up to 56 days.
* For Part 1, participants will stay at the study research center for 4 days after screening. There will be 2 other visits to the center to check on participants' health on Day 7 and Day 14.
* For Part 2, at 2 different times, participants will stay at the center for a period of 4 days at a time, after screening. There will be a break of about 7 days between stays. There will be 3 other visits to the center to check on their health on Day 7 (of each period) and on Day 14.
* For Part 3, participants will stay at the center for 17 days after screening. There will be 2 other visits to the center to check on their health on Day 21 and Day 28.

DETAILED DESCRIPTION:
The primary objective of the study is to evaluate the safety and tolerability of single and multiple ascending doses of BIIB145 in healthy adult participants.

The secondary objectives of the study are to evaluate the pharmacokinetics (PK) profile of single and multiple ascending doses of BIIB145 and its enantiomers in healthy adult participants; and the effect of food on the PK profile of BIIB145.

ELIGIBILITY:
Key Inclusion Criteria:

* Have a body mass index (BMI) between 18 and 32 kilograms per square metre (kg/m^2), inclusive, and a total body weight > 50 kilograms (kg) at Screening and Check-In.
* Must be in good health as determined by the Investigator, based on medical history and Screening evaluations. Good health is defined as no clinically relevant abnormalities identified by a detailed medical history, full physical examination, including blood pressure and pulse rate measurement, 12-lead electrocardiogram (ECG), and clinical laboratory tests.

Key Exclusion Criteria:

* History of any clinically significant blood disorders or cardiac, endocrine, gastrointestinal, hematologic, hepatic, immunologic, metabolic, urologic, pulmonary, neurologic, dermatologic, psychiatric, or renal disease, or other major disease, as determined by the Investigator.
* History of, or ongoing, malignant disease, including solid tumours and hematologic malignancies (except for basal cell carcinomas and squamous cell carcinomas that have been completely excised and considered cured at least 1 year prior to Check-In).
* History of uncontrolled bleeding, or any risk of bleeding that, in the opinion of the Investigator, is clinically significant.
* History of torsades de pointes or additional risk factors for torsades de pointes (e.g., heart failure, hypokalemia, or family history of long QT syndrome), in the opinion of the Investigator.
* Any values of coagulation parameters including international normalized ratio, prothrombin time, and activated partial thromboplastin time above upper limit of normal at Screening or Check-In.
* Systolic blood pressure > 150 millimetres of mercury (mmHg) or < 90 mmHg after resting for 5 minutes in the supine position at Screening and prior to dosing. If out of range, testing may be repeated once at Screening and once prior to dosing.
* Any live or attenuated immunization or vaccination given within 30 days prior to Check-In or planned to be given during the study period.
* Prior exposure to BIIB145 or any lymphocyte-depleting therapy or exposure to any lymphocyte-targeting therapy within 3 months prior to Check-In, or at least 5 half-lives or for the anticipated duration of the product's pharmacodynamics (PD) effects, whichever is longer.
* Known lumbar spine deformity, degenerative arthritis of the lumbar spine, history of lumbar spinal surgery, spinal infection, spinal mass or trauma, and/or known evidence on magnetic resonance imaging (MRI) contraindicating lumbar puncture (LP).

NOTE: Other protocol-defined Inclusion/Exclusion criteria may apply.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 104 (Estimated)
Dates: Start 2025-12-18 (Actual); Primary Completion 2027-02-02 (Estimated); Study Completion 2027-02-02 (Estimated)

PRIMARY OUTCOMES:
Parts A, B, and C: Number of Participants With Treatment Emergent Adverse Events (TEAEs) and Serious Adverse Events (SAEs) | Parts A and Part B: Up to Day 14; Part C: Up to Day 28
Parts A, B, and C: Number of Participants With Clinical Laboratory Abnormalities | Parts A and Part B: Up to Day 14; Part C: Up to Day 28
Parts A, B, and C: Number of Participants With Clinically Relevant Abnormalities in Vital Sign Parameters | Parts A and Part B: Up to Day 14; Part C: Up to Day 28
Part C: Number of Participants With Columbia Suicide Severity Rating Scale (C-SSRS) Events | Part C: Up to Day 28
Parts A, B, and C: Number of Participants With Potentially Clinically Relevant Abnormalities in 12-lead Electrocardiogram (ECG) Parameters | Parts A and B: Up to Day 14; Part C: Up to Day 28

SECONDARY OUTCOMES:
Parts A, B, and C: Area Under the Concentration-Time Curve (AUC) of BIIB145 | Pre-dose and at multiple timepoints post-dose (Parts A and B: Up to Day 4; Part C: Up to Day 17)
Parts A, B, and C: Maximum Observed Concentration (Cmax) of BIIB145 | Pre-dose and at multiple timepoints post-dose (Parts A and B: Up to Day 4; Part C: Up to Day 17)
Parts A, B, and C: Time to Maximum Observed Concentration (Tmax) of BIIB145 | Pre-dose and at multiple timepoints post-dose (Parts A and B: Up to Day 4; Part C: Up to Day 17)
Parts A, B, and C: Elimination Half-Life (t1/2) of BIIB145 | Pre-dose and at multiple timepoints post-dose (Parts A and B: Up to Day 4; Part C: Up to Day 17)
Parts A, B, and C: Apparent Clearance (CL/F) of BIIB145 | Pre-dose and at multiple timepoints post-dose (Parts A and B: Up to Day 4; Part C: Up to Day 17)
Parts A, B, and C: Apparent Volume of Distribution (Vz/F) of BIIB145 | Pre-dose and at multiple timepoints post-dose (Parts A and B: Up to Day 4; Part C: Up to Day 17)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Biogen
Locations (1):
- PPD Austin Clinic, Austin, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes
In accordance with Biogen's Clinical Trial Transparency and Data Sharing Policy on https://www.biogentrialtransparency.com/
URL: https://vivli.org/